CLINICAL TRIAL: NCT04180865
Title: The Dutch Parkinson and Cognition Study (DUPARC): A Prospective Study on Cognitive Pathology in de Novo Parkinson'Disease
Brief Title: The Dutch Parkinson and Cognition Study
Acronym: DUPARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Parkinson Platform Noord Nederland (Unknown)
Responsible Party: Principal Investigator, Teus van Laar, Professor of Neurology, University Medical Center Groningen
Other Study IDs: 201700171; NL60540.042.17 (Registry Identifier: Centrale Commissie Mensgebonden Onderzoek (CCMO))
Record Dates: First submitted 2019-11-04; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Treatment naive; Cognition; PET imaging; Acetylcholine; Magnetic Resonance Imaging; Ophthalmology; Gastrointestinal Microbiome; Neurodegenerative Diseases; Genetic subtyping
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces; Saliva; Plasma EDTA; Buffy coat (plasma EDTA); Serum;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: 150 de novo treatment naive Parkinson's disease patients.
- Healthy control subjects: 150 Healthy sex- and age-matched controls, also matched according to presence and severity of constipation, serving as a control group for microbiome composition analyses.

SUMMARY:
Parkinson Disease (PD) is a heterogeneous, progressive neurodegenerative disorder which is characterized by a variety of motor and non-motor symptoms. The DUPARC study is a single-centre longitudinal cohort study aimed at deeply phenotyping newly diagnosed PD patients. The main aim is to investigate the relationship between cognitive impairment and both cholinergic and dopaminergic neurodegeneration in the early stages of the disease. In addition, gastrointestinal and visual system dysfunction in PD and their role in the underlying pathology are further explored in a longitudinal setup. Treatment-naïve participants will undergo extensive motor- and non-motor assessment, imaging, and microbiome assessment at time of diagnosis, and will be followed for at least 3 years.

DETAILED DESCRIPTION:
Rationale:

Parkinson's disease (PD) is characterized by both motor and non-motor symptoms, including cognitive decline. Mild cognitive impairment (PD-MCI) is already present at time of diagnosis in 24-36% of PD patients. Cognitive impairment in PD is associated with both cholinergic and dopaminergic deficiencies in the brain. Although dopaminergic neuronal degeneration is quite well established in relationship to the motor impairment, the rate and extent of the cholinergic neuronal degeneration in the course of PD is unknown. It is also unclear how cholinergic and dopaminergic degeneration contributes to cognitive deficits found in early and more advanced PD and its role in the progression over time.

Objectives:

The primary objective is to establish the relationship between cognitive impairment and cholinergic neurodegeneration in de novo PD patients, by studying cholinergic imaging using [ 18 F]Fluoroethoxy-Benzovesamicol ([18F]FEOBV) positron emission tomography (PET) and neuropsychological performance over time.

Secondary objectives include: (1) the investigation of possible predictive factors using optical coherence tomography and (2) to determine the relative contributions of PD diagnosis and dopaminergic medication use to the changes in microbiota composition observed in PD patients.

Study design:

At baseline patients will undergo the following investigations and questionnaires: Demographics, detailed medical history, neuropsychological assessment, imaging including MRI brain, dopaminergic Fluoro-18-L-Dihydroxyphenylalanine (18F-FDOPA) and cholinergic FEOBV PET, optical coherence tomography (OCT) and microbiota composition. At one year follow-up subjects will undergo motor-, neuropsychological, and microbiota assessment. At 3 year follow up baseline measurements will be repeated in its entirety with the exception of the genetic and gastrointestinal assessments.

Study population:

150 de novo PD patients, recruited from the neurological practices in the northern area of the Netherlands and healthy control subjects. Healthy age-,sex- and constipation-matched controls will be assessed on microbiota composition

Assessment and endpoints related to gastroenterological assessment have been approved under a separate research protocol (NL61123.042.17 - CCMO) and has been officially linked to the overall protocol.

ELIGIBILITY:
Inclusion criteria

- Diagnosis Parkinson's disease

Exclusion criteria:

* The refusal to be informed about an unforeseen clinical finding.
* Dopaminergic medication use.

Exclusion from PET imaging:

* Pregnant women
* Breast feeding women

Exclusion from MRI:

* MRI incompatible implants in the body (e.g. prosthesis, pacemakers, implanted heart valves)
* Any risk of having metal particles in the eyes due to manual work without proper eye protections
* Tattoos containing red pigments that form a safety risk.

Exclusion from gastrointestinal assessment:

* Active or persistent primary disease of the gastrointestinal tract
* History of peritonitis, severe endometriosis, abdominal, intestinal or urogenital fistula,
* Hepatobiliary or pancreatic disease (except asymptomatic cholecystolithiasis)
* History of abdominal or anorectal surgery, except minor surgery such as uncomplicated appendectomy or cholecystectomy (>6 months ago).
* Severe gynaecological prolapse (grade III)
* Cancer and/or adjuvant treatment within the last 6 months
* Within the last three months: severe hypo- or hyperkalemia, narcosis, analgosedation, endoscopic procedure of the gastrointestinal tract, abdominal trauma
* Within the last three months: gastrointestinal tract infection, food intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 PD patients who are treatment naïve at baseline, diagnosed by a movement disorders specialist, based on the Movement Disorder Society Clinical Diagnostic Criteria for PD. Patients are recruited at partnering hospitals in the northern part of the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
[18F]FEOBV PET | Baseline
  Cortical and subcortical cholinergic innervation as measured by [18F] FEOBV PET imaging

SECONDARY OUTCOMES:
Cognitive screening | baseline
  General cognitive performance will be assessed using a cognitive screening; the Montreal Cognitive Assessment (MOCA). The MOCA test covers the important cognitive domains including memory, attention, executive function, language and visuospatial abilities, resulting in one total score of cognitive performance. MOCA score ranges between 0 and 30, with higher scores representing better performance.
Memory performance | baseline
  Memory performance will be calculated as an average Z-score of two cognitive tests; the Rey auditory verbal learning test for measuring verbal memory and the location learning test for measuring visual memory. Based on established normative data, a z-score for each test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from both tests will be averages to form one outcome measurement representing memory performance.
Attention and working memory performance | baseline
  Attention performance will be calculated as an average Z-score of three cognitive tests; the Stroop color-word test, the digit span and the Vienna test system reaction time measurement. Based on established normative data, a z-score for each test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from all three tests will be averages to form one outcome measurement representing attention performance.
Executive function performance | baseline
  Executive function performance will be calculated as an average Z-score of four cognitive tests; the trail making test, the Wisconsin card sorting test, the Hayling Sentence completion test and the letter fluency test. Based on established normative data, a z-score for each test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from all tests will be averages to form one outcome measurement representing executive performance.
Visouspatial abilities | baseline
  Cognitive visuospatial abilities will be calculated as an average Z-score of two cognitive tests; the Judgement of line orientation and the Map search subtest of the test of everyday attention. Based on established normative data, a z-score for each test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from all tests will be averages to form one outcome measurement representing visuospatial abilities.
Language performance | baseline
  Language performance will be calculated as an average Z-score of two cognitive tests; the Boston Naming test and the verbal fluency test. Based on established normative data, a z-score for each test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from all tests will be averages to form one outcome measurement representing language performance.
Social cognition | baseline
  Social cognition abilities will be represented as a z-score calculated from the performance on the FEEST; Facial Expression of Emotion Stimuli and tests. Based on established normative data, a z-score of the test outcome will be calculated, representing performance compared to an age-, gender- and educational level-matched control group. A Z-score of 0 (zero) represents a performance similar to the normative data. A positive z-score represents better performance, while a negative z-score represents worse performance. There is no minimum or maximum z-score. These z-scores from the FEEST test represents social cognition performance.
Brain grey matter volume | Baseline, 3 year follow-up
  Grey matter volume as measured by structural MRI.
resting state functional MRI | Baseline, 3 year follow-up
  resting state functional MRI
MRI: Arterial spin labeling | Baseline, 3 year follow-up
  cerebral blood perfusion as measured by arterial spin labeling MRI
MRI: Diffusion weighted image | Baseline, 3 year follow-up
  White matter assessment as measured by diffusion weighted image
MRI: susceptibility weighted image | Baseline, 3 year follow-up
  Brain hemorrhage and iron storage as measured by susceptibility weighted image
Optical Coherence tomography | Baseline and 3 year follow-up
  Imaging of the retinal cell layers
fecal zonulin | baseline
  fecal zonulin as one of the measures of intestinal wall permeability
Microbiota composition | Baseline and 1 year follow-up
  Taxonomic classification of gut microbiota composition based on 16s ribosomal RNA-gene sequencing.
fecal alpha1-antitrypsin | baseline
  fecal alpha1-antitrypsin as one of the measures of intestinal wall permeability
serum zonulin | baseline
  serum zonulin as one of the measures of intestinal wall permeability
serum lipopolysaccharide binding protein | baseline
  serum lipopolysaccharide binding protein as one of the measures of intestinal wall permeability
multi-sugar urinary excretion test | baseline
  multi-sugar urinary excretion test as one of the measures of intestinal wall permeability
Genetic subtyping | Baseline
  Saliva samples will be collected for clinical-genetic subtyping based on genome wide single-nucleotide polymorphism (SNP) analysis using the Illumina Screening Array (GSA-MD)
Movement Disorders Society Unified Parkinson's Disease Rating Scale III | Baseline, 1 year follow-up, 3 year follow-up
  Motor assessment measured by the Movement Disorders Society Unified Parkinson's Disease Rating Scale III, a scale describing motor performance specific for patients with Parkinson's disease. Score between 0 and 72, with a higher score indicating more severe motor impairment.
Change in [18F] FEOBV PET over 3 years | baseline, 3 year follow up
  Change in cortical and subcortical cholinergic innervation over a time period of 3 years, as measured by baseline and follow-up [18F] FEOBV

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire assessing anxiety and depression. Scores range from 0 to 42, with higher scores indicating more severe anxiety and depression symptoms
Utrechtse Coping Lijst | Baseline, 1 year follow-up, 3 year follow-up
  Dutch version of the Coping List; assessing coping style. The questionnaire consists of 47 items which can all be scored on a 1-4 scale and can be filled out by the participant. A higher score indicates a stronger involvement of that coping strategy.
The Dysexecutive Questionnaire | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire assessing dysexecutive problems in daily life. The DEX comprises of 20 items. All items are rates in terms of frequency on a 5-point scale: 0 (never), 1 (occasionally), 2 (sometimes), 3 (fairly often), 4 (very often). Scores are summed and the total scores range from 0 to 80, with higher scores indicating greater problems with executive functioning.
The Dutch Multifactor Fatigue Scale | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire assessing fatigue. The questionnaire consists of 38 items which can be rated on a 5-point scale. Scores are summed, with higher scores indicating more severe fatigue reported by the participant.
Questionnaire for Impulsive-Compulsive Disorder in Parkinson's Disease Rating Scale | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire for Impulsive-Compulsive Disorder in Parkinson's Disease Rating Scale (QUIP) is a questionnaire with 27 yes/no questions on impulsive-compulsive behavior. The total number of questions answered with "yes" is the main outcome measurement, with a higher score indicating more impulsive-compulsive symptoms.
Apathy Evaluation Scale | Baseline, 1 year follow-up, 3 year follow-up
  The Apathy Evaluation Scale (AES) is a questionnaire assessing apathy, comprised of 18 items, describing the subject's thoughts, feelings, and activity in the past 4 weeks. All items are rates in terms on a 4-point scale. Scores are summed and the total score ranges from 0 to 72, with higher scores indicating more severe presence of apathy symptoms
Movement disorders society - Non Motor Symptom Questionnaire; | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire assessing non-motor symptoms specific for patients with Parkinson's disease. The questionnaire consists of 30 yes/no questions on the occurrence of certain non-motor symptoms. The total number of questions answered with "yes" is used as outcome measure, indicating more presence of non-motor symptoms.
Rapid eye movement Sleep behavioral disorders (RBD) questionnaire | Baseline, 1 year follow-up, 3 year follow-up
  Questionnaire assessing Rapid eye movement (REM) sleep behavioral disorder. The questionnaire is a 10-item questionnaire with yes/no answers, of which question 6 consists of subitems. The number of questions answered with "yes" is considered the outcome measure, with a score ranging between 0 and 13. Higher scores indicate more REM sleep behavioral disorder symptoms.
Dietary assessment | Baseline, 1 year follow-up
  Dietary assessment. Participants are asked to complete a daily diary on their intake, including detailed description of what type of food/drinks, time of day and amount of intake for three consecutive days.
Stool frequency questionnaire | Baseline, 1 year follow-up
  Participants are asked to record their stool frequency for one week. Based on the questionnaire an average daily stoolfrequency is calculated and used as outcome measure.
Stool consistency questionnaire | Baseline, 1 year follow-up
  Stool consistency is recorded for one week by the patients using the Bristol Stool chart. The Bristol Stool chart is a 7 point rating scale with 1 representing separate hard lumps as stool consistency and 7 entirely liquid stool. An average is calculated representing average stool consistency for the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Teus van Laar, MD PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chrysou A, Heikka T, van der Zee S, Boertien JM, Jansonius NM, van Laar T. Reduced Thickness of the Retina in de novo Parkinson's Disease Shows A Distinct Pattern, Different from Glaucoma. J Parkinsons Dis. 2024;14(3):507-519. doi: 10.3233/JPD-223481. PMID 38517802
- [Derived] Boertien JM, van der Zee S, Chrysou A, Gerritsen MJJ, Jansonius NM, Spikman JM, van Laar T; PPNN Study Group. Study protocol of the DUtch PARkinson Cohort (DUPARC): a prospective, observational study of de novo Parkinson's disease patients for the identification and validation of biomarkers for Parkinson's disease subtypes, progression and pathophysiology. BMC Neurol. 2020 Jun 13;20(1):245. doi: 10.1186/s12883-020-01811-3. PMID 32534583